CLINICAL TRIAL: NCT01829490
Title: Phase I Trial to Evaluate the Safety and Immunogenicity of a ChAdOx1 85A Vaccination With and Without MVA85A Boost in Healthy BCG Vaccinated Adults
Brief Title: Safety Study of ChAdOx1 85A Vaccination With and Without MVA85A Boost in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TB034
Record Dates: First submitted 2013-03-26; First posted 2013-04-11 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Tuberculosis
Keywords: Vaccine; Immunogenicity
MeSH Terms: conditions — Tuberculosis | interventions — MVA 85A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Starter Group (Experimental): The first six volunteers will receive one dose of 5x10^9vp of ChAdOx1 85A intramuscular injection.
  Interventions: Biological: ChAdOx1 85A
- Group A (Experimental): 12 subjects will receive one dose of 2.5x10^10vp of ChAdOx1 85A intramuscular injection.
  Interventions: Biological: ChAdOx1 85A
- Group B (Experimental): 12 subjects will receive one dose of 2.5x10^10vp of ChAdOx1 85A by intramuscular injection, followed by a boost dose of 1x10^8pfu of MVA85A by intramuscular injection 56 days later.
  Interventions: Biological: ChAdOx1 85A; Biological: MVA85A
- Group C (Experimental): 12 subjects will receive two doses of 2.5x10^10vp of ChAdOx1 85A by intramuscular injection at day 0 and day 28, followed by a boost dose of 1x10^8pfu of MVA85A by intramuscular injection at day 119.
  Interventions: Biological: ChAdOx1 85A; Biological: MVA85A

INTERVENTIONS:
Biological: ChAdOx1 85A — Intramuscular injection
Biological: MVA85A — Intramuscular injection
  Arms: Group B; Group C

SUMMARY:
This is a Phase I trial to evaluate the safety and immunogenicity of a ChAdOx1 85A vaccination with and without MVA85A boost in healthy BCG vaccinated adults.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to enter the trial:

* Healthy adult aged 18-55 years
* Resident in or near Oxford (for CCVTM) or Birmingham (for WTCRF) and able to travel to Oxford for vaccinations for the duration of the trial period
* No relevant findings in medical history or on physical examination
* Confirmation of prior vaccination with BCG not less than 6 months prior to projected trial vaccination date (by visible BCG scar on examination or written documentation)
* Allow the Investigators to discuss the individual's medical history with their GP
* Use effective contraception for the duration of the trial period (females only)
* Refrain from blood donation during the trial
* Give written informed consent
* Allow the Investigator to register subject details with a confidential database to prevent concurrent entry into clinical trials
* Able and willing (in the Investigator's opinion) to comply with all the trial requirements

Exclusion Criteria:

Subjects must meet none of the following criteria to enter the trial:

* Laboratory evidence at screening of latent M. tb infection as indicated by a positive ELISpot response to ESAT6 or CFP10 antigens
* Clinical, radiological, or laboratory evidence of current active TB disease
* Shared a residence within one year prior to day 0 with an individual on anti-tuberculosis treatment or with culture- or smear-positive pulmonary tuberculosis
* Previous vaccination with any recombinant MVA, FP or adenoviral vector
* Clinically significant history of skin disorder, allergy, immunodeficiency (including HIV), cancer (except BCC or CIS), cardiovascular disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder, neurological illness, psychiatric disorder, drug or alcohol abuse
* History of serious psychiatric condition
* Concurrent oral or systemic steroid medication or the concurrent use of other immunosuppressive agents
* History of anaphylaxis to vaccination or any allergy likely to be exacerbated by any component of the trial vaccine including eggs
* Any abnormality of screening blood or urine tests that is deemed to be clinically significant or that may compromise the safety of the subject in the trial
* Positive HBsAg, HCV or HIV antibodies
* Female currently lactating, confirmed pregnancy or intention to become pregnant during trial period
* Use of an investigational medicinal product or non-registered drug, live vaccine, or medical device for 30 days prior to dosing with the trial vaccine, or planned use during the trial period
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned trial vaccination date
* Any other significant disease, disorder, or finding, which, in the opinion of the Investigator, may either put the subject at risk or may influence the result of the trial or may affect the subject's ability to participate in the trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2013-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Safety of ChAdOx1 85A vaccination with, and without, MVA85A boost vaccination in healthy, BCG vaccinated adults. | Six months following vaccination
  To evaluate the safety in healthy BCG-vaccinated subjects of ChAdOx1 85A vaccination, with and without MVA85A boost vaccination, by actively and passively collecting data on adverse events.

SECONDARY OUTCOMES:
To investigate the T-cell immune response of ChAdOx1 85A vaccination compared with ChAdOx1 85A vaccination with MVA85A boost vaccination. | Six months following vaccination
  To evaluate the systemic and mucosal cellular immunogenicity in healthy BCG-vaccinated subjects of ChAdOx1 85A vaccination, compared with ChAdOx1 85A vaccination with MVA85A boost vaccination, by comparing laboratory markers of cell mediated immunity in blood.

OTHER OUTCOMES:
To conduct further exploratory immunological analyses on samples from vaccinees in this trial. | Six months following vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Helen McShane, Principal Investigator — University of Oxford
Locations (2):
- United Kingdom (2):
  - Centre for Clinical Vaccinology and Tropical Medicine , University of Oxford, Oxford, Oxfordshire
  - The NIHR/ Wellcome Trust Clinical Research Facility, University of Birmingham, Birmingham, West Midlands

REFERENCES:
- [Derived] Crisan-Dabija R, Grigorescu C, Pavel CA, Artene B, Popa IV, Cernomaz A, Burlacu A. Tuberculosis and COVID-19: Lessons from the Past Viral Outbreaks and Possible Future Outcomes. Can Respir J. 2020 Sep 5;2020:1401053. doi: 10.1155/2020/1401053. eCollection 2020. PMID 32934758
- See also: Jenner Institute Clinical Trials — http://www.jenner.ac.uk/clinicaltrials